CLINICAL TRIAL: NCT03769766
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Curcumin to Prevent Progression of Biopsy Proven, Low-risk Localized Prostate Cancer Patients Undergoing Active Surveillance
Brief Title: Trial of Curcumin to Prevent Progression of Low-risk Prostate Cancer Under Active Surveillance
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, yair lotan, MD, Professor and Chief of Urologic Oncology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU 012018-071
Record Dates: First submitted 2018-12-05; First posted 2018-12-10 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; active surveillance; curcumin
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Curcumin; Sugars

STUDY DESIGN:
Intervention Model Description: placebo/active Curcumin
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Curcumin (Active Comparator): * Other names for the supplement: BCM-95 CG (Biocurcumax),Tumeric
  * Manufacture- DolCas Biotech, LLC.
  * Classification - type of agent: Supplement
  * Protocol dose: 500 mg twice
  Interventions: Drug: Curcumin
- Placebo (Placebo Comparator): Drug: placebo
  placebo orally twice a day Other Names: •sugar pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Curcumin — Take medication one 500 mg pill of BCM-95 taken twice daily
  Other Names: biocurcumax (BCM-95)
  Arms: Curcumin
Drug: Placebo — Take medication one 500mg pill twice daily
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
This is a prospective study to determine if the use of curcumin randomized against placebo will reduce cancer progression in patients with prostate cancer undergoing active surveillance.

DETAILED DESCRIPTION:
Prostate cancer is the most common cancer in men with an estimated 180,890 new cases and 26,120 deaths from prostate cancer expected in 2016 in the United States. Although the lifetime risk of developing prostate cancer, the risk of death is only about 3%. A major concern regarding the utility of prostate cancer screening is the risk of over diagnosis and subsequent overtreatment. Many patients with small low grade cancers might not benefit from treatment and treatment can result in lower quality of life. A major concern for patients and physicians using active surveillance (AS) is the risk for progression of disease. Several reviews of active surveillance suggest that stage or grade progression occur in approximately 30% of patients with some patients choosing treatment due to anxiety. Overall survival in AS series is uniformly high but the need for close monitoring and anxiety associated with risk of progression has inhibited use among patients.

There are no currently accepted medications to reduce risk of progression in patients with active surveillance. With the rising use of AS, there is a role for therapies to reduce risk for progression in this population. One promising source of therapies involves use of nutraceuticals for the prevention and treatment of human diseases. Curcumin is a widely studied nutraceutical that was first discovered about two centuries ago from the rhizomes of Curcuma longa (turmeric). Curcumin is a safe supplement and in this study we will evaluate if it reduces risk of cancer progression compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40-89 years
* Biopsy proven, low-risk, localized prostate cancer (minimum of 8 cores)
* May have had biopsy within last 12 months
* ≤4 separate locations in the prostate involved with cancer. If multiple cores are obtained from same lesion or area than this will count as one location.
* Gleason score ≤6 with no Gleason pattern 4
* Clinical stage T1c-T2a/b
* Serum PSA ≤15 ng/ml
* Life expectancy > 5 years

Exclusion Criteria:

* Any previous prostate cancer treatment (radiotherapy, chemotherapy, hormonal therapy, oral glucocorticoids, GnRH analogues, prostatectomy)
* Concurrent or previous use within 6 months of screening of any 5α-reductase inhibitor
* Use of anabolic steroids or drugs with antiandrogenic properties
* Prostate volume >150 cm³
* Patients who are taking antiplatelet, anticoagulant agents or have a history of a bleeding disorder. Patients taking 81 mg of Aspirin will be allowed to enroll with close observation
* History of gastric or duodenal ulcers or untreated hyperacidity syndromes. Patients on stable doses (2 months of therapy) of GERD medication allowed.
* Patients who are currently taking Curcumin and are unwilling to stop or plan to take Curcumin during the study
* Patients with a history of gallbladder problems or gallstones or biliary obstruction, unless patient had cholecystectomy

Ages: 40 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients have to have prostate cancer
Enrollment: 291 (Estimated)
Dates: Start 2019-03-11 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
The primary end point is rate of disease progression. | 2 years
  The primary endpoint is the number of patients who have progressed at 2 years of follow up defined as one of the following events: receipt of primary therapy for prostate cancer (eg, prostatectomy, radiation, hormonal therapy) or pathologic progression (> 4 cores involved, ≥ 50% of any core involved, or any Gleason score ≥ 7)

CONTACTS AND LOCATIONS:
Overall Officials: Yair Lotan, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States